CLINICAL TRIAL: NCT02594592
Title: Combined Assessment of the Osteoporosis Self-assessment Tool for Asians and the One-Minute Osteoporosis Risk Test in a Wuhan Population
Brief Title: Clinical Value of Self-assessment Risk of Osteoporosis in Chinese
Status: Completed | Type: Observational
Sponsor: Hongmei Zhang (Other)
Responsible Party: Sponsor-Investigator, Hongmei Zhang, director of department of endocrinology, Wuhan Integrated Traditional Chinese and Western Medicine Hospital
Organization: Wuhan Integrated Traditional Chinese and Western Medicine Hospital (Other)
Other Study IDs: WuhanITCWMH
Record Dates: First submitted 2015-10-19; First posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Osteoporosis Self-Assessment Tool; One-Minute Osteoporosis Risk Test; Asians
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Younger Women: Younger Women (age ≤ 55 years),complete questionaire
  Interventions: Other: questionaire
- Younger Men: Younger Men (age ≤ 55 years),complete questionaire
  Interventions: Other: questionaire
- Older Men: Older Men (age > 55 years). complete questionaire
  Interventions: Other: questionaire
- Older Women: Older Women (age > 55 years),complete questionaire
  Interventions: Other: questionaire

INTERVENTIONS:
Other: questionaire — Arm: Experimental :questionaire medium risk, and high risk.(more than one positive answer about questionaire) Arm:Active Comparator: questionaire low risk (none of positive answer about questionaire)

SUMMARY:
This cross-sectional study aimed to validate the effectiveness of the combined use of the Osteoporosis Self-Assessment Tool for Asians (OSTA) and the One-Minute Osteoporosis Risk Test (IOF test) in a population from Wuhan, China.

DETAILED DESCRIPTION:
This cross-sectional study was a field investigation. A total of 400 Wuhan residents who visited the Health Examination Department at our hospital were invited to participate in this study. Potential participants were informed of the aim and procedures and were asked to sign an informed consent form before participation. Inclusion criteria were as follows: age of at least 20 years, able to read and fill out the questionnaire, and willingness to participate. Exclusion criteria were as follows: severe liver, heart, or kidney impairment, and tumor. Procedures of the study were in accordance with the Declaration of Helsinki and were approved by the local ethics committee.

The study population was divided into four groups according to age and sex: Younger Women (age ≤ 55 years), Younger Men (age ≤ 55 years), Older Women (age > 55 years), and Older Men (age > 55 years). A research assistant and a nurse distributed the Chinese version of the IOF test to participants. The Chinese version of the IOF test includes 10 questions, two of which are specific to women and one to men. The maximum number of risk factors is 8 for women and 9 for men. Individuals were regarded as susceptible to osteoporosis risk if they answered "yes" to any of the 10 questions.

To assess the grade of osteoporosis risk, the OSTA index was calculated by the equation (body weight (kg) - age (years))*0.2. An OSTA index of -1 to -4 is regarded as medium risk, greater than -1 as low risk, and less than -4 as high risk.

ELIGIBILITY:
Inclusion Criteria:

* age of at least 20 years, able to read and fill out the questionnaire, and willingness to participate.

Exclusion Criteria:

* severe liver, heart, or kidney impairment, and tumor. Procedures of the study were in accordance with the Declaration of Helsinki and were approved by the local ethics committee.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: age of at least 20 years, able to read and fill out the questionnaire, and willingness to participate.
Sampling Method: Probability Sample
Enrollment: 389 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
validate the effectiveness of the combined use of the Osteoporosis Self-Assessment Tool for Asians and the One-Minute Osteoporosis Risk Test | 1 day
  The IOF test were filled out by participants. The Chinese version of the IOF test includes 10 questions, two of which are specific to women and one to men. The maximum number of risk factors is 8 for women and 9 for men. Individuals were regarded as susceptible to osteoporosis risk if they answered "yes" to any of the 10 questions.The OSTA index was calculated by the equation (body weight (kg) - age (years))*0.2. weight in kilograms. age in years.An OSTA index of -1 to -4 is regarded as medium risk, greater than -1 as low risk, and less than -4 as high risk. Then detect any association between the results of IOF test and the risk grade.